CLINICAL TRIAL: NCT00981734
Title: Effects of a Hiking Study About the Functional Autonomy Levels in Old Women Analyzed by the Family Health Program
Brief Title: Hiking Improves the Functional Autonomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Camilo Castelo Branco (Other)
Responsible Party: Rubens Ceasr Lucena da Cunha, Universidade Castelo Branco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 0042/2008
Record Dates: First submitted 2009-09-14; First posted 2009-09-22 (Estimated); Last update posted 2009-09-22 (Estimated); Status verified 2009-09

CONDITIONS: Aging
Keywords: Aging; functionality; life style; To have more than sixty years
MeSH Terms: interventions — CHE protein, Arabidopsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Hiking — Three times by a week, thirty minutes, controlling heart frequency between fifty five per cent and seventy five per cent.
  Other Names: Funcionality, life style.

SUMMARY:
This is an experimental research study. The subjects were randomized into two groups: Experimental group (EG; n=58, age: 67 ± 6 old) and Control group (CG; n=40; age: 70 ± 6 old). All were physically active without strictly obeying in regularity of the program of physical activity.

The functional autonomy was evaluated by the amount of tests of Group Development of Latin American Maturity (GDLAM). It consists of hiking ten meters (C10m); standing up from the sitting position (SSP); to stand up from the ventral decubitus position (SSPVD); to stand up from a chair and be able to walk around your home (SCWH); and to be able to wear and remove a t-shirt (DTS). These tests have showed similar results in indice of GDLAM (IG). The intervention took place three times a week, with intensity that has varied between fifty five to seventy five per cent of the frequency maximum from heart.

DETAILED DESCRIPTION:
In the physical evaluation, the participants were asked that they bathe with clothes (swimsuit, trunks) to measure the body composition, stature and IMC. All of the results were recorded in elaborated cards by the researcher.

The participants were physically evaluated through systemic observation during 16 weeks. The first collection of data occurred in the first week of April and the second collection occurred in the first week of August, 2009 during the morning.

A weighing machine with the unit of Filizola registered to INMETRO (precision of 100 grams) was used to evaluate body composition. Stature was measured through the use of a Estadiometer registered to INMETRO (precision of 1 mm). In order to evaluate the functional autonomy, GDLAM (Group Development of Latin American Maturity) created by Dantas and Vale, was used. It consists of hiking ten meters (C10m); standing up from the sitting position (SSP); to stand up from the ventral decubitus position (SSPVD); to stand up from a chair and be able to walk around your home (SCWH); and to be able to wear and remove a t-shirt (DTS). Everybody was measured in seconds and consists of a score called the General Indice of the GDLAM (IG).

The results of reference for classification of the functional autonomy level were the same for IG and its components and GDLAM. The intervention took place three times per week (Monday, Wednesday, Friday) from 5 PM to 5:45 PM. Intensity varied between 50% and 75% of the frequency maximum from heart (FMH) obtained by the equation: FMH = 220 - age. The FMH was controlled by the standardization of the heart frequency (HF) from the carotid at six seconds and then multiplied by ten. This HF WAS measured by the participants themselves. They received training and orientations to learn the right method.

All the participants had their HF measured by monitors, at least one time per session. Therefore after the self-standardization, with the aim to confirm the identified results by the older women. The moment of standardization of the HF varied due to the voice of the responsible teacher or asked by the monitor close to the old woman.

The sessions were spread out in the subsequent ways:

* Warm up: Duration five to ten minutes of articular exercises of upper body, neck, trunk and lower body.
* Development: twenty to thirty minutes of hiking in a natural method.
* To came back to calmness: three to five minutes of sitting elongated and/or laying down: neck, upper and lower body and trunk; using the changed method by segment. The activity of intervention was oriented at a controlled environment as the surface (plain and does not glide) and markation of the walked distances (field jogging does not count - 260 meters) where the training was controlled by the time of hiking, according to Norms of the American College Sport of Medicine and of the fifth Brazilian Norm of arterial Hypertension, that has the requirement of a minimum frequency of three times per week with the duration of twenty and thirty minutes; adequate to have a good mean to physiological adaptations in etary group.

Statistic Evaluation:

Descriptive Statistics were used with average, error-standard, median, standard deviation, minimum and maximum and absolute delt. The normality of the sample was evaluated by the test by Shapiro-Wilk (GC) and by Kolmogorov Smirnov (GE). To analyze the answer variables, comparisons were made between groups, t-student test couplet or by Wilcoxon, when appropriate (homogeneous or heterogenous distributions of the data, respectively). To make evaluations between groups the parametric test by ANOVA was used in two ways, followed by Post Hoc de Scheffe. The study used the level of p < 0.05 to test the statistical significance. The results were evaluated by Excel and the Statistical Package for the Social Science® (SPSS), version 14.0.

ELIGIBILITY:
Inclusion Criteria:

* Registered in a program of family health (PFH),
* Age above 60 years,
* Hypertension,
* Not be trainee of physical activity and those who were at clinical conditions that composed the research.

Exclusion Criteria:

* Old women with any kind of infirmity that could interferes in study or that becomes a factor of prevention of the tests that were designed for functional anatomy.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2008-09; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
10 meters | seconds

SECONDARY OUTCOMES:
meters | seconds

CONTACTS AND LOCATIONS:
Overall Officials: Functional Autonomy older women, Principal Investigator — Universidade Camilo Castelo Branco
Locations (1):
- Rubens Cesar Lucena da Cunha, Juazeiro do Norte, Ceará, Brazil